CLINICAL TRIAL: NCT04109014
Title: Depression, Meth Use, and Safe Sex Behaviors: Assessing the Feasibility and Acceptability of an HIV Cognitive Behavioral Intervention for Young Adult Latina Women
Brief Title: FASTLANE II: Reducing Sex, Drug, and Mental Health Risk
Acronym: FLII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Alice Cepeda, Associate Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UP-15-00628
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Methamphetamine Abuse; HIV/AIDS; Depression; Sex, Unsafe
Keywords: Cognitive Behavioral; Qualitative Interviews; Motivational Interviewing
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Depression; Unsafe Sex

STUDY DESIGN:
Intervention Model Description: Quasiexperimental, single group pretest-posttest study design and qualitative interviews to evaluate feasibility, acceptability and effect.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FASTLANE II Group (Other): Participants will participate in the FASTLANE II Intervention. Counseling sessions will focus on: 1) depressive symptoms, 2) methamphetamine use, and 3) sexual risk behaviors. Three sessions will be devoted to each topic area. Trained staff will use a client-centered approach and develop a goal for each area alongside the participant. Counseling sessions will remain confidential and will not be audio recorded.
  Interventions: Other: FASTLANE II

INTERVENTIONS:
Other: FASTLANE II — The intervention will consist of nine weekly hour-long individual counseling sessions. The FL II sessions utilize a combination of Cognitive Behavioral Therapy (CBT) and Motivational Interviewing (MI) to reduce sexual risk behaviors and mental health symptoms. Thus, individuals develop a "toolbox" for mood self-management to improve emotional self-regulation and reduce maladaptive coping mechanisms to minimize drug and sex risk behavior. Participants will be considered as completing the FASTLANE Intervention upon completion of the nine weeks of sessions.

SUMMARY:
The study uses a repeated measures, single group pretest-posttest design methodology to examine the feasibility, acceptability, and preliminary effectiveness of the FASTLANE II intervention aimed at decreasing risky sex behaviors among active methamphetamine using women. The study's methodology consists of two phases: 1) The feasibility and evaluation of recruitment capability and intervention effectiveness, and 2) qualitative acceptability interviews.

DETAILED DESCRIPTION:
Specific Aims Methamphetamine use among young adult Latina women with histories of intimate partner violence are at disproportionate risk for Human Immunodeficiency Virus (HIV) and sexually transmitted infection (STI). Studies demonstrate that these women are also at extremely high risk for a myriad of mental health conditions, including depression. There is promising support that addressing the co-occurrence of drug use and depression can lead to increased safe sex behaviors, positive outcomes and HIV/STI risk reduction. However, there are countless systemic barriers to engaging drug using young adult women who face high rates of psychological, interpersonal relationship and legal problems into safe sex interventions.

In response to the University of Southern California (USC) Clinical and Translational Science Institute (CTSI) Clinical and Community Research Award, this application proposes to assess the feasibility of an integrated HIV behavioral intervention, FASTLANE II that has preliminary evidence of efficacy in increasing safer sex behaviors and simultaneously targeting depressive symptoms among active drug users. FASTLANE II utilizes cognitive behavioral therapy (CBT) and incorporates motivational interviewing (MI) techniques as well as central theoretical components from the theory of reasoned action. The study will deliver FASTLANE II for a new population and new setting and obtain initial data on its feasibility, acceptability and preliminary outcome data. Specifically, the proposed application builds upon an on-going National Institute on Drug Abuse (NIDA) funded R01, "Proyecto San Antonio Latina Trajectory Outcomes (SALTO) - 5R01DA039269-04, a longitudinal community-based study examining long-term health outcomes of drug and partner violence victimization trajectories for a cohort of Mexican American women in San Antonio, Texas (SAT). Findings demonstrate a high-needs population with high rates of STIs, illicit drug use and depression confounded by low rates of access and utilization of health care. The investigators will employ a quasi- experimental, single group pretest-posttest study design and qualitative interviews to evaluate feasibility, acceptability and effect. Specifically, the investigators plan to pursue the following specific aims:

1. To assess the feasibility of recruiting and retaining active methamphetamine using Mexican American women in SAT;
2. Obtain outcome data (depression, sex risk and methamphetamine use) for a new population in a new setting;
3. Explore participant's perceptions of the acceptability of the FASTLANE II intervention.

This study will provide preliminary data that would inform a future randomized controlled trial (RCT) to implement a promising HIV intervention for this underserved vulnerable population using National Institute of Health (NIH) Funding Opportunity Announcement Number PAR-17-490/ PAR-17-491 "Implementing the Most Successful Interventions to Improve HIV/AIDS Outcomes in US Communities". Moreover, the study takes advantage of a unique team of collaborators including: 1) the University of Incarnate Ward San Antonio; 2) the University of California San Diego and 3) the University of Southern California.

Research Strategy Significance Research has demonstrated the heightened risk for HIV/STI infection among methamphetamine users engaged in unprotected sexual behaviors. Studies demonstrate significantly more sex partners, engagement in anal sex behavior, engagement in prostitution or exchange of sex for drugs and less likely to use condoms. Despite this, few interventions exists to increase safer sex behaviors among populations of methamphetamine users. This is particularly important given that curtailing and/or changing drug use behaviors is a time-intensive specialized process and often times not a realistic goal for active users engaged in sexual risk behaviors. Thus, the proposed study will add to the limited interventions that exist in reducing sexual risks in the context of active drug (methamphetamine) using women.

Our study population represents one of the largest and fastest growing Hispanic subgroup in the U.S. living in poverty (27% compared to 15% U.S. general population). Mexican Americans' disadvantaged status (e.g. high poverty and declining economic progress and educational attainment) has been shown to persist with each succeeding (i.e. 3rd and 4th) generation. Confounding this status is evidence documenting intimate partner violence (IPV) and related substance use and sexual risk patterns among women. There are important limitations in the existing knowledge resulting from a lack of attention to Mexican Americans in studies of women's health and from issues related to the lack of attention to the barriers that contribute to underutilization of healthcare services. This study will contribute to examining the feasibility and acceptability of an intervention that takes into account drug using women's unique susceptibility for mental health conditions and engaging in sexual risk behaviors. While it is particularly important to recognize the sociocultural disadvantage these women experience, there is an immediate need to address the acute vulnerability that heightens their risk on a day-to-day basis.

The proposed study builds off emerging findings from "Proyecto SALTO" that demonstrate a current rate of 56% that tested positive for Herpes Simplex Virus Type 2 (HSV-2) infection and strong comorbidity with drug use, Hepatitis C, sexual violence, incarceration, and mental illness. Moreover, preliminary results from the parent study demonstrate a high-needs population of methamphetamine users with high rates of co-occurring risky sex behavior and detrimental mental health.

Approach

Quasi-Experimental Design and Methods

Study Setting - San Antonio

The San Antonio population is more than 1 million, of which more than 50% is of Mexican descent. SAT is among the top 10 cities with the largest number of people living in distressed zip codes and has the highest level of spatial inequality between zip codes. Building upon the research team's "Proyecto SALTO", the proposed intervention study site is located in the most distressed zip code. Findings demonstrate a marginalized and vulnerable population of young women with high rates of STIs, illicit drug use, and depression confounded by low rates of access and utilization of healthcare.

Community Advisory Board (CAB). A CAB will be assembled to advise the research team. The investigators will take advantage of the existing CAB members for the ongoing SAT NIDA funded study who have expressed their willingness to provide insights and suggestions for the implementation of the intervention. It will meet three times to advise and discuss such issues as cultural norms, values and beliefs, attitudes towards methamphetamine use, gender sensitivity, sexual behavior cultural scripts, etc. The CAB will monitor progress of the project and provide guidance on both cultural and community issues that develop during the course of the study.

Phase I: Feasibility and Evaluation of Recruitment Capability The objective for aim 1 is to evaluate the feasibility of recruitment and retention of appropriate participants. The investigators intend to recruit 40 participants through a variety of methods including a) existing participants in the ongoing "Proyecto SALTO" study; b) street outreach in targeted neighborhoods; and c) snowball sampling techniques. The investigators will assess and document participant flow through recruitment rates, eligibility criteria, and resulting sample characteristics in order to evaluate the feasibility of FASTLANE II in this setting. The investigators will also assess adherence rates to study procedures, intervention attendance, and engagement. In order to minimize underreporting of sensitive behavior, the investigators will utilize REDCAP for data collection purposes. Computerized assessments will occur at baseline, posttest and 4 months post-baseline. Participants will be compensated $30 for completing study assessments.

FASTLANE II (FL II) Intervention Developed by our University of California, San Diego (UCSD) collaborator (Patterson), FL II counseling sessions are highly interconnected given they are built on multiple frameworks. For instance, self-efficacy and outcome expectancies are developed through Social Cognitive Theory (SCT) and intention is explored through the Theory of Reasoned Action (TRA). While MI teaches individuals to use existing skills in risky situations,

CBT compliments the therapy by building on existing strategies and knowledge in order to develop new approaches individuals can use to improve mood and reduce risk behavior. Thus, individuals develop a "toolbox" for mood self-management to improve emotional self-regulation and reduce maladaptive coping mechanisms to minimize drug and sex risk behavior. The intervention consists of nine weekly face-to-face (i.e., individual) counseling sessions, focused on addressing the following: 1) depressive symptoms, 2) methamphetamine use, and 3) sexual risk behavior. Counselors use a client-centered approach and develop a goal for each area alongside the participant. Three sessions are devoted to each described elsewhere.

Results from the FL II intervention among a sample of randomized HIV-negative, heterosexual methamphetamine users found reductions in depression, meth use, and condom-less sex. Limited efficacy was demonstrated in changes over time that pointed towards gender moderation effects. That is, FL II demonstrates the importance in interventions targeting gender-specific factors, in particular for women who demonstrate unique vulnerabilities (homelessness, gendered power dynamics, dependent children, lower income, more severe trading sex for meth).

Analysis -Analyses will focus on the proportion of participants who complete the intervention and retention at 4- month follow-up. The investigators will use χ2 tests (or Fisher's exact tests if cell sizes are small) for categorical and t-tests for continuous variables to explore whether participant attributes are associated with intervention and study completion. χ2 tests will explore change from baseline to 4-month follow-up on the categorical outcome variables. Paired sample t-tests will be used to examine whether there was change on the outcomes from baseline to follow-up. The qualitative analysis will implement 4 inductive strategies. 1) Item level: unrestricted line-by-line reading and initial coding for items and/or elements. 2) Pattern level: more focused coding to establish linkages among classifications. 3) Structural level: organizes relationships among patterns of the data into larger sociocultural constructs. 4) Interpretation: provides meaning of structures in relation to existing content and used to assist in adaptation of intervention.

Limitations - A problem that could arise is that the investigators are unable to recruit the proposed sample. Given the team's highly successful work, trust and rapport with young adult women in "Proyecto SALTO", the investigators are confident that this would not occur. However, should this occur, the investigators will implement direct advertising recruitment using bulletin board posts/flyers at local community- based organizations working with targeted population.

ELIGIBILITY:
Inclusion Criteria:

* Resident of San Antonio, Texas
* Female
* Mexican-American
* HIV-negative
* 18 years of age or older
* Self-identify as heterosexual
* Have had unprotected sex with at least one opposite sex partner during the previous 2 months
* Indicate that they have snorted or smoked methamphetamine at least once during the previous 2 months

Exclusion Criteria:

* Not a resident of San Antonio, Texas
* Male
* Not Mexican-American
* HIV-positive
* Younger than 18 years of age
* Do not self-identify as heterosexual
* Have not had unprotected sex with at least one opposite sex partner during the previous 2 months
* Indicate that they have not snorted or smoked methamphetamine at least once during the previous 2 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Depression | 9-12 weeks
  Participants will be asked to complete the Beck Depression Inventory (BDI-II) scale. A total of 21 items assess depressive symptoms over the past 2 weeks (including today), and are summed to create a summary score (alpha = 0.91). We used established cutoffs for minimal (0-13), mild (14-19), moderate (20-28), and severe depressive symptoms (29-63).
Sex Practices | 9-12 weeks
  Assesses number of times participants engaged in sexual behavior, (vaginal, oral, and anal sex). Follow-up questions assess number of times these sexual acts were protected. Use of condoms or oral dams or nonpenetrative (e.g., manual sex) excluding oral sex. Using these data, three outcome variables will be used: (a) total protected sex acts, (b) total unprotected sex acts, and (c) percentage of safer sex behaviors (i.e., ratio) by dividing protected sex behaviors by the total number of sex behaviors over the past 2 months.
Negotiating Self-Efficacy for Safer Sex | 9-12 weeks
  Seven questions pertaining to self-efficacy for negotiation of safer sex, including perceived ability to bring up the topic of safer sex with any partner, negotiate condom use with any partner, and convince a partner to use a condom if he or she resisted. Participants presented with a statement about being able to negotiate safer sex (e.g., ''I can persuade partners to try different types of condoms'') and rate agreement ranging from 1 (strongly disagree) to 4 (strongly agree). Total sum score with higher scores greater self-efficacy.
Methamphetamine Use | 9-12 weeks
  Asked to report number of days and grams (or preferred unit) of methamphetamine used in the past 30 days. They will be asked how often they snort, smoked, injected, injected in combination with another drug, or used in any other way in the past 2 months. Response options 0 = never, 1 = once in a while, 2 = fairly often, and 3 = very often. The items will be summed to create a summary score of "frequency of meth use across different methods in the past 2 months." Amount responses will be converted to grams using a standard formula (e.g., 8 ball ¼ 3.5 g; ounce ¼ 28 g). Converted values will be multiplied by number of times used to calculate the number of grams of methamphetamine used in the past 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Cepeda, PhD, Principal Investigator — University of Southern California
Locations (1):
- Proyecto SALTO Office, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rigby SW, Johnson LF. The relationship between intimate partner violence and HIV: A model-based evaluation. Infect Dis Model. 2017 Feb 16;2(1):71-89. doi: 10.1016/j.idm.2017.02.002. eCollection 2017 Feb. PMID 29928730
- [Background] Ulibarri MD, Strathdee SA, Patterson TL. Sexual and drug use behaviors associated with HIV and other sexually transmitted infections among female sex workers in the Mexico-US border region. Curr Opin Psychiatry. 2010 May;23(3):215-20. doi: 10.1097/YCO.0b013e32833864d5. PMID 20308903
- [Background] Zlotnick C, Johnson DM, Kohn R. Intimate partner violence and long-term psychosocial functioning in a national sample of American women. J Interpers Violence. 2006 Feb;21(2):262-75. doi: 10.1177/0886260505282564. PMID 16368765
- [Background] Bonomi AE, Anderson ML, Cannon EA, Slesnick N, Rodriguez MA. Intimate partner violence in Latina and non-Latina women. Am J Prev Med. 2009 Jan;36(1):43-48. doi: 10.1016/j.amepre.2008.09.027. PMID 19095164
- [Background] Ulibarri MD, Hiller SP, Lozada R, Rangel MG, Stockman JK, Silverman JG, Ojeda VD. Prevalence and characteristics of abuse experiences and depression symptoms among injection drug-using female sex workers in Mexico. J Environ Public Health. 2013;2013:631479. doi: 10.1155/2013/631479. Epub 2013 May 12. PMID 23737808
- [Background] Mausbach BT, Semple SJ, Strathdee SA, Zians J, Patterson TL. Efficacy of a behavioral intervention for increasing safer sex behaviors in HIV-positive MSM methamphetamine users: results from the EDGE study. Drug Alcohol Depend. 2007 Mar 16;87(2-3):249-57. doi: 10.1016/j.drugalcdep.2006.08.026. Epub 2006 Dec 19. PMID 17182196
- [Background] Zule WA, Costenbader EC, Meyer WJ Jr, Wechsberg WM. Methamphetamine use and risky sexual behaviors during heterosexual encounters. Sex Transm Dis. 2007 Sep;34(9):689-94. doi: 10.1097/01.olq.0000260949.35304.22. PMID 17471112
- [Background] McCoy HV, McCoy CB, Lai S. Effectiveness of HIV interventions among women drug users. Women Health. 1998;27(1-2):49-66. doi: 10.1300/J013v27n01_04. PMID 9640634
- [Background] Ennis, S., M. Rios-Vargas, & N.G. Albert, The Hispanic Population 2010. 2011.
- [Background] Motel, S.E.P., Hispanics of Mexican Origin in the United States, 2010. 2012, Pew Research Center.
- [Background] Telles, E.E.V.O., Generations of Exclusion: Mexican Americans, Assimilation, and Race. 2008, Russell Sage Foundation.
- [Background] Caetano R, Field CA, Ramisetty-Mikler S, McGrath C. The 5-year course of intimate partner violence among White, Black, and Hispanic couples in the United States. J Interpers Violence. 2005 Sep;20(9):1039-57. doi: 10.1177/0886260505277783. PMID 16051726
- [Background] Smith CA, Ireland TO, Park A, Elwyn L, Thornberry TP. Intergenerational continuities and discontinuities in intimate partner violence: a two-generational prospective study. J Interpers Violence. 2011 Dec;26(18):3720-52. doi: 10.1177/0886260511403751. Epub 2011 Aug 1. PMID 21810795
- [Background] Jennings WG, Reingle JM, Staras SA, Maldonado-Molina MM. Substance Use as a Risk Factor for Intimate Partner Violence Overlap: Generational Differences Among Hispanic Young Adults. Int Crim Justice Rev. 2012 Jun 1;22(2):139-152. doi: 10.1177/1057567712442943. PMID 25125930
- [Background] Nowotny KM, Frankeberger J, Rodriguez VE, Valdez A, Cepeda A. Behavioral, Psychological, Gender, and Health Service Correlates to Herpes Simplex Virus Type 2 Infection among Young Adult Mexican-American Women Living in a Disadvantaged Community. Behav Med. 2019 Jan-Mar;45(1):52-61. doi: 10.1080/08964289.2018.1447906. Epub 2018 May 9. PMID 29558260
- [Background] United States Census Bureau, DP-1-Profile of General Population and Housing Characteristics: 2010. 2010.
- [Background] Economic Innovation Group, The 2016 Distressed Communities Index: An Analysis of Community Well- Being Across the United States. Economic Innovation Group.
- [Background] Quinn SC. Ethics in public health research: protecting human subjects: the role of community advisory boards. Am J Public Health. 2004 Jun;94(6):918-22. doi: 10.2105/ajph.94.6.918. PMID 15249289
- [Background] Pitpitan, E.V., et al., Cognitive behavioral therapy for HIV-negative heterosexual meth users: the FASTLANE II intervention. Cognitive and Behavioral Practice, 2014. 21(2): p. 176-190.
- [Background] Pitpitan EV, Semple SJ, Zians J, Strathdee SA, Patterson TL. Mood, Meth, Condom Use, and Gender: Latent Growth Curve Modeling Results from a Randomized Trial. AIDS Behav. 2018 Sep;22(9):2815-2829. doi: 10.1007/s10461-018-2147-9. PMID 29754267
- [Background] Beck, A., R. Steer, and G. Brown, Manual for the BDI-II. 1996, San Antonio, TX: Psychological Corporation.
- [Background] Corbin, J.M. and A. Strauss, Grounded theory research: Procedures, canons, and evaluative criteria. Qualitative sociology, 1990. 13(1): p. 3-21.
- [Background] Glaser, B. and A. Strauss, Discovery of grounded theory: Strategies for qualitative review. 1967, Chicago, IL: Aldine De Gruyter.
- [Background] LeCompte, M.D. and J.J. Schensul, Analyzing & interpreting ethnographic data. 1999: Rowman Altamira.
- [Background] Ragin, C.C., The Comparative Method: Moving Beyond Qualitative and Quantitative Strategies. 1987, Los Angeles: University of California Press.
- [Background] Ragin CC. Using qualitative comparative analysis to study causal complexity. Health Serv Res. 1999 Dec;34(5 Pt 2):1225-39. No abstract available. PMID 10591281
- [Background] Spradley, J., The Ethnographic Interview. New York, NY: Holt, Rinehart and Winston. Inc, 1979.